CLINICAL TRIAL: NCT01839019
Title: Safety, Tolerability and Pharmacokinetics of Single Escalating Doses of ODM-102: A Randomised, Double-blind, Placebo-controlled, Single Centre Study in Healthy Males
Brief Title: Safety and Tolerability Study With Single Ascending Doses of ODM-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3099003
Record Dates: First submitted 2013-04-17; First posted 2013-04-24 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Each subject will receive 2 single doses of study drug, either both of them active doses or the other placebo.
  Interventions: Drug: Placebo for ODM-102
- ODM-102 (Experimental): Each subject will receive 2 single doses of study drug, either both of them active doses or the other placebo.
  Interventions: Drug: ODM-102

INTERVENTIONS:
Drug: ODM-102 — Single dose escalation
  Arms: ODM-102
Drug: Placebo for ODM-102 — Single dose escalation
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of escalating single doses of ODM-102 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history and physical examination.
* Finnish-speaking males between 18 and 45 years of age (inclusive).
* Body mass index (BMI) between 18.0-30.5 kg/m2 (inclusive).
* Weight 55.0-100.0 kg (inclusive).

Exclusion Criteria:

* Suspected poor compliance or inability to communicate well with the investigator.
* Veins unsuitable for repeated venipuncture.
* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastro-intestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
* Any condition requiring regular concomitant drug treatment, including herbal products, or likely to need any concomitant drug treatment during the study.
* Susceptibility to severe allergic reactions.
* Intake of any medication that could affect the outcome of the study within 2 weeks prior to the first study drug administration or within less than 5 times the elimination half-life of the medication.
* Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
* Inability to refrain from using nicotine-containing products during the stay in the study centre.
* Inability to refrain from consuming caffeine-containing beverages during the first 24 hours after treatment administration e.g. propensity to experience headache when abstaining from caffeine-containing beverages.
* Blood donation or loss of a significant amount of blood within 2 months prior to the screening visit.
* Abnormal 12-lead ECG finding of clinical relevance after 10 min rest in supine position at the screening visit
* HR < 45 beats/minute or > 90 beats/minute after 10 minutes rest in supine position at the screening visit.
* At the screening visit, systolic BP < 90 mmHg or > 140 mmHg after 10 minutes in supine position, diastolic BP < 50 mmHg or > 90 mmHg after 10 minutes in supine position, or symptomatic orthostatic hypotension, or decrease of ≥ 20 mmHg of systolic BP or decrease of ≥ 10 mmHg of diastolic BP after 3 minutes in standing position.
* Abnormal 24-hour Holter ECG recording of possible or confirmed clinical relevance
* Any abnormal laboratory value, vital sign, or physical examination finding, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk to the subject if he takes part in the study.
* Suspected current use of illicit drugs (according to medical history enquiry or physical examination), positive drug screen or history of long-term drug abuse.
* Positive serology to human immunodeficiency virus antigen/antibodies (HIVAgAb), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibodies (HCVAb).
* Participation in another clinical drug study within 3 months prior to the first treatment administration in this study.
* Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the subject.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety measures, i.e. assessing adverse events, vital signs, ECG and safety laboratory values | about a month

SECONDARY OUTCOMES:
Pharmacokinetics | 5 days per period
  Explore the PK profile (e.g. Cmax, tmax, AUC, t1/2), screen circulating metabolites and determine protein binding.

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, Principal Investigator — Clinical Research Services Turku, CRST
Locations (1):
- Clinical Research Services Turku, CRST, Turku, Finland